CLINICAL TRIAL: NCT03071679
Title: A Randomized, Evaluator-blinded, Vehicle-controlled Study to Explore the Pharmacodynamic Effects of Omiganan and Omiganan in Combination With Imiquimod in Healthy Volunteers
Brief Title: Topical Challenge With Omiganan and Imiquimod in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Other
Other Study IDs: CLS001-CO-PR-015; 2016-004702-34 (EudraCT Number)
Record Dates: First submitted 2017-02-21; First posted 2017-03-07 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Healthy
MeSH Terms: interventions — Omiganan; Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Omiganan (Experimental)
  Interventions: Drug: Omiganan
- Imiquimod (Experimental)
  Interventions: Drug: Imiquimod
- Omiganan 1% and Imiquimod (Experimental)
  Interventions: Drug: Omiganan 1% and Imiquimod
- Omiganan 2.5% and Imiquimod (Experimental)
  Interventions: Drug: Omiganan 2.5% and Imiquimod
- Placebo (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omiganan — Omignan 1%, 2.5%
  Arms: Omiganan
Drug: Imiquimod — Imiquimod 15mg
  Arms: Imiquimod
Drug: Omiganan 1% and Imiquimod — Omiganan 1% and Imiquimod
  Arms: Omiganan 1% and Imiquimod
Drug: Omiganan 2.5% and Imiquimod — Omiganan 2.5% and Imiquimod
  Arms: Omiganan 2.5% and Imiquimod
Drug: Placebo — Vehicle
  Arms: Placebo

SUMMARY:
This study has a randomized, evaluator-blinded, vehicle- controlled study to assess the pharmacodynamics of omiganan and omiganan with imiquimod in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 45 years of age, inclusive. Healthy status is defined by absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, haematology, blood chemistry, blood serology and urinalysis.
* Body mass index (BMI) between 18 and 30 kg/m2, inclusive, and with a minimum weight of 50 kg.
* Fitzpatrick skin type I-III (Caucasian)
* Subjects and their partners of childbearing potential must use effective contraception, for the duration of the study and for 3 months after the last dose.
* Able and willing to give written informed consent and to comply with the study restrictions.

Exclusion Criteria:

* Any disease associated with immune system impairment, including auto-immune diseases, HIV and transplantation patients
* Family history of psoriasis
* History of pathological scar formation (keloid, hypertrophic scar)
* Have any current and / or recurrent pathologically, clinical significant skin condition.
* Previous use of imiquimod/ resiquimod/ gardiquimod
* Known hypersensitivity to the (non)investigational drug, drugs of the same class, or any of their excipients.
* Hypersensitivity for dermatological marker at screening
* Requirement of immunosuppressive or immunomodulatory medication within 30 days prior to enrollment or planned to use during the course of the study.
* Use of topical medication (prescription or over-the-counter [OTC]) within 30 days of study drug administration, or less than 5 half-lives (whichever is longer) in local treatment area
* Tanning due to sunbathing, excessive sun exposure or a tanning booth within 3 weeks of enrollment.
* Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year.
* Loss or donation of blood over 500 mL within three months (males) or four months (females) prior to screening
* Pregnant, a positive pregnancy test, intending to become pregnant, or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Clinical Evaluation | 6 Days
  Erythema grading scale
Pharmacodynamic (Biomarkers) | Within 2 Weeks
  Local biomarker sequencing
Pharmacodynamic (Histology) | Within 2 Weeks
  Histological parameters assessment
Pharmacodynamic (Immunohistochemistry) | Within 2 Weeks
  Identification of lymphocytes and lineage cells
Pharmacodynamic (TAP) | Within 6 Days
  Qualitatively and Quantitatively analyze biomarkers captured by Trans Epidermal Patch (TAP)
pharmacodynamic (LSCI) | Within 6 Days
  Assess cutaneous microcirculation using laster speckle imager
Pharmacodynamic (Colorimetry) | Within 6 Days
  Colorimetric assessment by erythema grading scale
Pharmacodynamic (Photography) | Within 2 Weeks
  Photographs of treatment sites will be taken
Pharmacodynamic (Thermography) | Within 2 Weeks
  Skin temperature measurements will be taken

SECONDARY OUTCOMES:
Local tolerability | 2 Weeks
  Visual Analogue Scale (NRS) pruritus and pain
Safety (AE) | 2 Weeks
  Adverse Events will be collected throughout the study
Safety (Vital Signs) | 2 Weeks
  Vital Signs will be collected throughout the study
Safety (Laboratory Safety Testing) | 2 Weeks
  Lab samples collected in various timepoints within the study
Safety (ECG) | Within 3 Weeks
  ECGs will be collected before beginning and end of study

CONTACTS AND LOCATIONS:
Overall Officials: J. (Koos) Burggraaf, MD, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- LUMC/Centre for Human Drug Research, Leiden, Netherlands